CLINICAL TRIAL: NCT04155879
Title: Atrial Fibrillation Recurrence Following Cardioversion: the Role of Clinical Factors and Alpha Defensin Levels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HYMC-19-0074
Record Dates: First submitted 2019-09-11; First posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Colchicine; Electric Countershock

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Investigator and participants will be blinded regarding levels of anti-inflammatory markers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Cardioversion without treatment with Colchicine
- Treatment group (Active Comparator): This arm will undergo cardioversion followed by Colchicine (0.5 mg 2x per day) for six months
  Interventions: Drug: Colchicine Tablets; Procedure: Cardioversion

INTERVENTIONS:
Drug: Colchicine Tablets — Administration of Colchicine at a dose of 0.5mg 2x a day for six months.
  Arms: Treatment group
Procedure: Cardioversion — Electrical or pharmacologic restoration of sinus rhythm
  Arms: Treatment group

SUMMARY:
Atrial fibrillation and inflammation are strongly correlated. The aim of this study is to evaluate whether inflammation markers (alpha Defensin) predict maintenance of sinus rhythm following cardioversion. A secondary aim is to evaluate the role of Colchicine, an anti-inflammatory medication, in reducing the recurrence rate of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation
* Candidate for cardioversion

Exclusion Criteria:

* Colchicine allergy
* Hepatic or renal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial fibrillation | 12 months
  Atrial fibrillation recurrence rates over the next 12 months will be determined based on medical records and ECG documentation between treatment group (Colchicine) and control group.

SECONDARY OUTCOMES:
Alpha Defensin levels in patients with recurrence of atrial fibrillation | 12 months
  Alpha Defensin levels will be measured in patients with recurrence of atrial fibrillation and compared to levels in patients without recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No